CLINICAL TRIAL: NCT04110847
Title: Traditional Chinese Medicine Formula in the Treatment of Osteoarthritis of Knees or Hips. A Randomized Double-Blind, Placebo-Controlled Clinical Trial.
Brief Title: Traditional Chinese Medicine Formula in the Treatment of Osteoarthritis of Knees or Hips.
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Chung Shan Medical University (Other)
Responsible Party: Principal Investigator, Cheng-Chung Wei, Professor, Chung Shan Medical University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Basic Science
Other Study IDs: CS09165
Record Dates: First submitted 2019-09-30; First posted 2019-10-01 (Actual); Last update posted 2019-10-01 (Actual); Status verified 2019-09

CONDITIONS: Osteoarthritis
MeSH Terms: conditions — Osteoarthritis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- TCM OA1 (Active Comparator): JING CEIH SHERN YUAN EXTRACT PILL "CHUANG SONG ZONG" 3 TABLET For 2 Times per day
  Interventions: Drug: JING CEIH SHERN YUAN EXTRACT PILL
- Placebo (Placebo Comparator): Placebo 3 TABLET For 2 Times per day
  Interventions: Drug: JING CEIH SHERN YUAN EXTRACT PILL

INTERVENTIONS:
Drug: JING CEIH SHERN YUAN EXTRACT PILL — Oral use, 3#BID

SUMMARY:
To investigate the efficacy and safety of OA1 Extract capsules in the treatment of patients with knee or hip osteoarthritis (OA).

DETAILED DESCRIPTION:
This trial was a 12 weeks' randomized, double-blind, placebo-controlled study. The study was approved by the Institutional Review Board of Chung Shan Medical University hospital, and signed informed consent was obtained from each patient. Sixty patients of osteoarthritis of knees or hips were enrolled in this study. Inclusion criteria were: age 20 to 80 years; primary osteoarthritis in at least 1 knee or hip, verified; at least moderate pain during 2 weeks before random assignment to treatment, as identified by the Western Ontario and McMaster Universities (WOMAC) LK3.0 Osteoarthritis Index pain subscale for more than 4.

Primary outcome measures were WOMAC at week 12.

Secondary outcome measures were WOMAC at week 4 and 8; Visual analogue scale (VAS) , Quality of life by SF-36, patient global assessment (PGA), at week 4, 8 and 12; serum levels of osteocalcin, C-terminal telopeptide(CTX), Hs-CRP, and ESR.

ELIGIBILITY:
Inclusion Criteria:

* 1. Age ≥20 years old 2. Written informed consent obtained 3. Been diagnosed with knee or hip osteoarthritis 4. The physician interpretation of X-ray identification and joint space narrowing or bone spurs confirmed 5. In randomized trials before entering if used steroids or non-steroid medications osteoarthritis stable doses required at least one week 6. The WOMAC osteoarthritis index of the degree of pain assessment in the past two weeks at least> 4ppm pain

Exclusion Criteria:

* 1. Pregnant or breast-feeding women. 2. Chemotherapy or radiation therapy in cancer patients

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2010-03-22 (Actual); Primary Completion 2011-12-05 (Actual); Study Completion 2012-01-10 (Actual)

PRIMARY OUTCOMES:
Western Ontario and McMaster Universities (WOMAC) | week 0, week 12
  The investigators use WOMAC to compared the difference between the week 12 and week 0

SECONDARY OUTCOMES:
serum osteocalcin level | week 0, week 12
  The investigators use serum osteocalcin level to compared the difference between week 12 and week 0
serum C-terminal telopeptide (CTX) level | week 0, week 12
  The investigators use serum CTX level to compared the difference between week 12 and week 0
Western Ontario and McMaster Universities (WOMAC) | week 0, week 4, week 8
  The investigators use WOMAC to compared the difference between the week 4 and week 0, week 8 and week 0
Visual Analog Scale for pain (VAS) | week 0, week 4, week 8, week 12
  The investigators use VAS to compared the difference between the week 4 and week 0, week 8 and week 0, week 12 and week 0
Physicians Global Assessment to measure quality of life (PGA) | week 0, week 4, week 8, week 12
  The investigators use PGA to compared the difference between the week 4 and week 0, week 8 and week 0, week 12 and week 0
Quality of life by SF-36 | week 0, week 4, week 8, week 12
  The investigators use SF-36 to compared the difference between the week 4 and week 0, week 8 and week 0, week 12 and week 0
High sensitivity C-reactive protein (Hs-CRP) | week 0, week 12
  The investigators use Hs-CRP to compared the difference between the week 12 and week 0
Erythrocyte sedimentation rate (ESR) | week 0, week 12
  The investigators use ESR to compared the difference between the week 12 and week 0

CONTACTS AND LOCATIONS:
Overall Officials: Cheng Ching Wei, Ph. D., Study Director — Chung Shan Medical University

IPD SHARING:
Plan to Share IPD: No